CLINICAL TRIAL: NCT05946083
Title: The Brain, the Bug, and the Binge: a Double-blind, Randomized Controlled Trial Investigating the Interplay Between Binge Drinking, Gut Microbiota and Brain Functioning
Brief Title: The Brain, the Bug, and the Binge: the Interplay Between Binge Drinking, Gut Microbiota, and Brain Functioning
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minho (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Eduardo López-Caneda, Assistant Reseacher, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CEICSH 078/2022; PTDC/PSI-ESP/1243/2021 (Other Grant/Funding Number: Portuguese Foundation for Science and Technology)
Record Dates: First submitted 2023-06-15; First posted 2023-07-14 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Binge Drinking
Keywords: Adolescence; Young Adulthood; Alcohol; Binge Drinking; Gut Microbiome; Microbiota-Gut-Brain Axis; Magnetic Resonance Imaging; Pro-inflammatory cytokines; Psychobiotics; Randomized Controlled Trial
MeSH Terms: conditions — Binge Drinking

STUDY DESIGN:
Intervention Model Description: Binge Drinkers will be randomly distributed for one of two groups: 23 subjects with inulin intervention and 23 subjects with maltodextrin intervention (~50 % male and ~50 % female in each group).
  There will also be a non-interventional control group consisting of 36 non/low-drinkers.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Binge Drinkers with Inulin Intervention (Active Comparator): 23 binge drinkers (~50 % male and ~50 % female) will be given a daily dose of inulin.
  Interventions: Dietary Supplement: Inulin Intervention
- Binge Drinkers with Maltodextrin Intervention (Placebo Comparator): 23 binge drinkers (~50 % male and ~50 % female) will be given a daily dose of maltodextrin.
  Interventions: Dietary Supplement: Maltodextrin Intervention
- Non/Low-Drinkers (No Intervention): 36 non/low-drinkers will not be given any dietary fiber.

INTERVENTIONS:
Dietary Supplement: Inulin Intervention — For 6 weeks, 23 binge drinkers will be given a daily dose (divided into three times a day) of 15g of a dietary fiber with benefits for intestinal bacteria (inulin).
  Arms: Binge Drinkers with Inulin Intervention
Dietary Supplement: Maltodextrin Intervention — For 6 weeks, 23 binge drinkers will be given a daily dose (divided into three times a day) of 15g of dietary fiber with no specific benefits for the intestinal microbiome (maltodextrin).
  Arms: Binge Drinkers with Maltodextrin Intervention

SUMMARY:
Adolescence and youth are periods of significant maturational changes which seems to involve greater susceptibility to disruptive events in the brain such as binge drinking (BD). This prevalent pattern of consumption -characterized by repeated alcohol intoxications- is of special concern, as it has been associated with major neurocognitive impairments in the young brain.

Recent studies indicate that alcohol may disrupt the gut microbiota (GM) and that these disruptions may lead to impairments in brain and behavior. Also, interventions with psychobiotics have been shown to result in reductions in alcohol-induced damage and in improvements on cognitive and brain functioning.

Thus, the present proposal will explore the effects of BD on GM. Additionally, a GM intervention with psychobiotics both in-vivo and in-vitro, will determine whether improvements in GM composition/function may lead to reductions of alcohol-induced brain damage in BD-population, a barely unexplored research field with major clinical applications.

DETAILED DESCRIPTION:
The present study protocol aims to determine the interaction between alcohol consumption, brain function and gut microbiota through several levels of analysis, including techniques to measure brain activity (i.e., magnetic resonance imaging), paradigms to measure cognitive performance, collection of stool and blood samples, and questionnaires. Additionally, this study will investigate the relationship between alcohol, brain activity and gut microbiota and how this can be modified through our diet. The sample will be composed by a cohort of young college students (18-23 years) from the University of Minho (UM; Braga, Portugal) selected according to their drinking patterns. Eighty-two participants will be recruited from UM: 36 non/low-drinkers and 46 binge drinkers (BDs) matched for age and gender. Recruitment will be carried out through an online survey broadcasted using the institutional email. This survey will include a simple sociodemographic section and items regarding the use of alcohol (Alcohol Use Disorder Identification Test - AUDIT, frequency of alcohol consumption, number of drinks consumed on each day of the past week, speed of drinking, etc.). After sample selection, participants will be submitted to the following steps: (1) clinical interview - addresses questions relating to psychological, medical, personal and family history, including questions related to history of alcohol and drug use and some specific questionnaires relating to substance use, as well as those related to physical and psychological symptoms, and personality; (2) neuroimaging assessment - will consist of a structural and functional magnetic resonance imaging (fMRI) at the Hospital de Guimarães (Portugal), while performing different cognitive tasks; (3) evaluation of some microorganisms residing in the gut and certain inflammatory markers - each participant will be asked to collect stool and blood samples; (4) evaluation of the potential of an intervention with psychobiotics.

Thus, this protocol involves the following phases:

1. pre-intervention, consisting of the assessment of the variables of interest to the study by means of a clinical interview, neuropsychological testing, collection of stool and blood samples, and MRI recordings.
2. intervention (only for BDs), consisting of taking a prebiotic for 6 weeks. Depending on the group to which they will be allocated, the participant will take one of two types of fiber: a fiber with benefits for intestinal bacteria (inulin) or a similar fiber with no specific benefits for the intestinal microbiome (maltodextrin). Each participant will not know which group they belong to in order not to bias the results of the study according to scientific standards.
3. post-intervention, which will consist in the re-assessment of the variables previously assessed in the pre-intervention phase.
4. follow-up, consisting of the assessment and monitoring of levels of alcohol consumption and craving during the 3 months following the intervention phase.

ELIGIBILITY:
Inclusion Criteria:

* College students whose native language is Portuguese;
* Age 18-23 years;
* Binge Drinkers: report (i) drinking 4 (for women)/5 (for men) or more drinks on one occasion at least once a month, (ii) drinking at a speed of at least two drinks per hour during these episodes (which brings blood alcohol concentration to 0.08 g/dL or above), and (iii) having an AUDIT score < 20.
* Non/Low-Drinkers: report (i) never drinking 4/5 or more drinks on one occasion and (ii) having an AUDIT score ≤ 4.

Exclusion Criteria:

* Use of illicit drugs as determined by the Drug Use Disorders Identification Test (DUDIT);
* Alcohol abuse (i.e., AUDIT ≥ 20);
* Personal history of psychopathological disorders (according to DSM-V criteria);
* History of traumatic brain injury or neurological disorder;
* Family history (mother/father) of alcoholism diagnosis of substance abuse;
* Occurrence of one or more episodes of loss of consciousness for more than 30 minutes;
* Non-corrected sensory deficits;
* Diagnosis of any gut disease/problems or other medical conditions: inflammatory bowel disease, irritable bowel syndrome, Crohn's Disease, celiac disease, lactose intolerance, autoimmune disease;
* Consumption of medical drugs with psychoactive effects (e.g., antidepressants, anxiolytics or benzodiazepines) during the 4 weeks prior to the experiment;
* Use of any of the following drugs in the last 4 weeks: laxatives, antibiotics, anticoagulants, non-steroidal anti-inflammatory drugs, analgesics, corticosteroids;
* No type of metal object implanted in the body, especially in the head (orthodontic appliances are not excluded).

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Fecal Microbiota - Species Richness | At baseline (pre-intervention)
  Faecal samples will be collected from all participants for microbiota α-diversity analysis by 16S rRNA metagenomics (Illumina sequencing). The Chao1 Index will be used as an estimator of nonparametric microbial species richness in each sample.
Fecal Microbiota - Species Richness | Immediately post-intervention.
  Faecal samples will be collected only from binge drinkers subjected to the intervention for microbiota α-diversity analysis by 16S rRNA metagenomics (Illumina sequencing). The Chao1 Index will be used as an estimator of nonparametric microbial species richness in each sample.
Fecal Microbiota - Species Diversity | At baseline (pre-intervention)
  Faecal samples will be collected from all participants for microbiota α-diversity analysis by 16S rRNA metagenomics (Illumina sequencing). The Shannon Diversity Index (metric combining richness and evenness, with equal weighting given to abundant and rare species) and the Simpson Diversity Index (metric of richness and evenness, in which more weighting is given to abundant species) will be used.
Fecal Microbiota - Species Diversity | Immediately post-intervention
  Faecal samples will be collected only from binge drinkers subjected to the intervention for microbiota α-diversity analysis by 16S rRNA metagenomics (Illumina sequencing). The Shannon Diversity Index (metric combining richness and evenness, with equal weighting given to abundant and rare species) and the Simpson Diversity Index (metric of richness and evenness, in which more weighting is given to abundant species) will be used.
Fecal Microbiota - Quantification of SCFAs levels | At baseline (pre-intervention)
  The concentration of short-chain fatty acids (SCFAs) present in each collected faecal sample shall be quantified by High Performance Liquid Chromatography (HPLC).
Fecal Microbiota - Quantification of SCFAs levels | Immediately post-intervention.
  The concentration of SCFAs present in each collected faecal sample shall be quantified by HPLC.

SECONDARY OUTCOMES:
Alcohol Consumption - Drinking pattern | Immediately post-intervention
  The AUDIT will be administered to characterize the drinking pattern of the participants. AUDIT scores ≤ 4 reveal low risk of alcohol use; scores between 5 and 20 represent excessive alcohol consumption; and scores ≥ 20 indicate very high risk for alcohol dependence and warrant further diagnostic evaluation for alcohol dependence.
Alcohol Consumption - Drinking pattern | 3 months post-intervention
  The AUDIT will be administered to characterize the drinking pattern of the participants. AUDIT scores ≤ 4 reveal low risk of alcohol use; scores between 5 and 20 represent excessive alcohol consumption; and scores ≥ 20 indicate very high risk for alcohol dependence and warrant further diagnostic evaluation for alcohol dependence.
Alcohol Craving - Short-term acute craving | Immediately post-intervention
  Short-term alcohol craving levels will be assessed using the ACQ-SF-R at the present moment. Total minimum score: 1 (low level of alcohol craving); Total maximum score: 7 (high level of alcohol craving).
Alcohol Craving - Short-term acute craving | 3 months post-intervention
  Short-term alcohol craving levels will be assessed using the ACQ-SF-R at the present moment. Total minimum score: 1 (low level of alcohol craving); Total maximum score: 7 (high level of alcohol craving).
Neuropsychological Evaluation - Memory | At baseline (pre-intervention)
  The Delayed Matching to Sample (DMS) from Cambridge Neuropsychological Test Automated Battery (CANTAB) will be used to assess both simultaneous visual matching ability and short-term visual recognition memory, for non-verbalisable patterns.
Neuropsychological Evaluation - Memory | Immediately post-intervention
  The Delayed Matching to Sample (DMS) from Cambridge Neuropsychological Test Automated Battery (CANTAB) will be used to assess both simultaneous visual matching ability and short-term visual recognition memory, for non-verbalisable patterns.
Neuropsychological Evaluation - Emotion and Social Cognition | At baseline (pre-intervention)
  The Emotion Recognition Task (ERT) from CANTAB will measure the ability to identify six basic emotions (sadness, happiness, fear, anger, disgust, and surprise) in facial expressions along a continuum of expression magnitude.
Neuropsychological Evaluation - Emotion and Social Cognition | Immediately post-intervention
  The Emotion Recognition Task (ERT) from CANTAB will measure the ability to identify six basic emotions (sadness, happiness, fear, anger, disgust, and surprise) in facial expressions along a continuum of expression magnitude.
Neuropsychological Evaluation - Executive Function | At baseline (pre-intervention)
  The performance of the cognitive domain comprising high-level thinking and decision-making will be assessed through CANTAB, namely the Cambridge Gambling Task (CGT, to assess decision-making and risk behaviour outside a learning context), Intra-Extra Dimensional Set Shift (IED, to assess cognitive flexibility), Spatial Working Memory (SWM, to identify working memory strategies and errors) and Stop Signal Task (SST, to measure response inhibition/impulse control).
Neuropsychological Evaluation - Executive Function | Immediately post-intervention
  The performance of the cognitive domain comprising high-level thinking and decision-making will be assessed through CANTAB, namely the Cambridge Gambling Task (CGT, to assess decision-making and risk behaviour outside a learning context), Intra-Extra Dimensional Set Shift (IED, to assess cognitive flexibility), Spatial Working Memory (SWM, to identify working memory strategies and errors) and Stop Signal Task (SST, to measure response inhibition/impulse control).
Alcohol Cue Reactivity - Emotional measures | At baseline (pre-intervention)
  The reactivity to alcoholic cues will be assessed using the Alcohol Cue Reactivity (ACR) task. The full task includes a total of 80 trials with 40 alcoholic and 40 non-alcoholic images obtained from the Amsterdam Beverage Picture Set. The emotional responses for each image in terms of valence and arousal task, will be registered using the Self-Assessment Manikin (valence: from 1 = "very unpleasant" to 9 ="very pleasant"; arousal: from 1 = "not arousing" to 9 = "highly arousing") during the ACR task.
Alcohol Cue Reactivity - Emotional measures | Immediately post-intervention.
  The reactivity to alcoholic cues will be assessed using the ACR task. The full task includes a total of 80 trials with 40 alcoholic and 40 non-alcoholic images obtained from the Amsterdam Beverage Picture Set. The emotional responses for each image in terms of valence and arousal task, will be registered using the Self-Assessment Manikin (valence: from 1 = "very unpleasant" to 9 ="very pleasant"; arousal: from 1 = "not arousing" to 9 = "highly arousing") during the ACR task.
Memory Inhibition Performance | At baseline (pre-intervention)
  Memory Inhibition (MI), specifically alcohol-related MI, will be assessed using the Think/No-Think Alcohol (TNTA) task. Percentage of correct responses (for Think, No-Think and Baseline items) in the TNTA task will be computed according to the following formula: ((number of correctly recalled items)/(number of previously learned items))×100. Correct responses correspond to the items learned during the learning phase and correctly recalled during the memory test phase.
Memory Inhibition Performance | Immediately post-intervention.
  MI, specifically alcohol-related MI, will be assessed using the TNTA task. Percentage of correct responses (for Think, No-Think and Baseline items) in the TNTA task will be computed according to the following formula: ((number of correctly recalled items)/(number of previously learned items))×100. Correct responses correspond to the items learned during the learning phase and correctly recalled during the memory test phase.
Ability of Emotional Recognition | At baseline (pre-intervention)
  Emotional recognition capacity will be assessed through the Emotion Discrimination (ED) task. ED assesses the brain's preconscious and conscious responses to emotional faces. The complete task includes a total of 120 images of human faces (60 men and 60 women), showing the main negative emotions: angry, sadness and fear.
Ability of Emotional Recognition | Immediately post-intervention.
  Emotional recognition capacity will be assessed through the ED task. ED assesses the brain's preconscious and conscious responses to emotional faces. The complete task includes a total of 120 images of human faces (60 men and 60 women), showing the main negative emotions: angry, sadness and fear.
Blood samples - Presence of Inflammatory Markers | At baseline (pre-intervention)
  Blood samples will be collected from all participants. The presence and abundance of the following cytokines will be analyzed: Tumour Necrosis Factor α (TNF-α) and Interleukins (IL-1β, IL-6, IL-10).
Blood samples - Presence of Inflammatory Markers | Immediately post-intervention.
  Blood samples will be collected only from binge drinkers subjected to the intervention. The presence and abundance of the following cytokines will be analyzed: Tumour Necrosis Factor α (TNF-α) and Interleukins (IL-1β, IL-6, IL-10).
Neurofunctional level - Think/No-Think Alcohol (TNTA) Task | At baseline (pre-intervention)
  The TNTA task assesses memory inhibition mechanisms in alcohol-related contexts. It involves three phases - Learning, Think/No-Think and Memory Test - during which participants memorise pairs of images (human faces with a neutral expression and alcoholic/non-alcoholic beverages) and are subsequently instructed to actively recall or suppress these associations.
Neurofunctional level - Think/No-Think Alcohol (TNTA) Task | Immediately post-intervention
  The TNTA task assesses memory inhibition mechanisms in alcohol-related contexts. It involves three phases - Learning, Think/No-Think and Memory Test - during which participants memorise pairs of images (human faces with a neutral expression and alcoholic/non-alcoholic beverages) and are subsequently instructed to actively recall or suppress these associations.
Neurofunctional level - Emotional Face Matching (EFM) Task | At baseline (pre-intervention)
  The EFM task assesses emotional recognition ability and pre-conscious and conscious neural responses to emotional faces and geometric forms. During each trial, participants view three emotional faces or shapes (one on top and two on the bottom, in a triangular configuration) and are instructed to identify the emotion/shape at the top of the screen and match it with the corresponding one at the bottom using handheld response buttons.
Neurofunctional level - Emotional Face Matching (EFM) Task | Immediately post-intervention
  The EFM task assesses emotional recognition ability and pre-conscious and conscious neural responses to emotional faces and geometric forms. During each trial, participants view three emotional faces or shapes (one on top and two on the bottom, in a triangular configuration) and are instructed to identify the emotion/shape at the top of the screen and match it with the corresponding one at the bottom using handheld response buttons.
Neurofunctional level - Alcohol Cue Reactivity (ACR) Task | At baseline (pre-intervention)
  The ACR task assesses the emotional and attentional response to alcoholic stimuli. Participants are shown images of alcoholic and non-alcoholic drinks, interspersed with oddball blocks containing neutral objects, to which they must respond by pressing a button. After viewing all images, participants are asked to rate their emotional responses to the alcoholic or non-alcoholic beverage images in terms of valence, arousal, and desire.
Neurofunctional level - Alcohol Cue Reactivity (ACR) Task | Immediately post-intervention
  The ACR task assesses the emotional and attentional response to alcoholic stimuli. Participants are shown images of alcoholic and non-alcoholic drinks, interspersed with oddball blocks containing neutral objects, to which they must respond by pressing a button. After viewing all images, participants are asked to rate their emotional responses to the alcoholic or non-alcoholic beverage images in terms of valence, arousal, and desire.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo G. López-Caneda, PhD, Principal Investigator — Psychological Neuroscience Laboratory, Psychology Research Center, University of Minho, Portugal.
Locations (1):
- Psychological Neuroscience Laboratory, Psychology Research Center, University of Minho, Braga, Gualtar, Braga, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carbia C, Bastiaanssen TFS, Iannone LF, Garcia-Cabrerizo R, Boscaini S, Berding K, Strain CR, Clarke G, Stanton C, Dinan TG, Cryan JF. The Microbiome-Gut-Brain axis regulates social cognition & craving in young binge drinkers. EBioMedicine. 2023 Mar;89:104442. doi: 10.1016/j.ebiom.2023.104442. Epub 2023 Feb 2. PMID 36739238
- [Background] Sousa SS, Sampaio A, Marques P, Lopez-Caneda E, Goncalves OF, Crego A. Functional and structural connectivity of the executive control network in college binge drinkers. Addict Behav. 2019 Dec;99:106009. doi: 10.1016/j.addbeh.2019.05.033. Epub 2019 Jun 3. PMID 31487578
- [Background] Almeida-Antunes N, Crego A, Carbia C, Sousa SS, Rodrigues R, Sampaio A, Lopez-Caneda E. Electroencephalographic signatures of the binge drinking pattern during adolescence and young adulthood: A PRISMA-driven systematic review. Neuroimage Clin. 2021;29:102537. doi: 10.1016/j.nicl.2020.102537. Epub 2020 Dec 17. PMID 33418172
- [Background] White A, Hingson R. The burden of alcohol use: excessive alcohol consumption and related consequences among college students. Alcohol Res. 2013;35(2):201-18. doi: 10.35946/arcr.v35.2.11. PMID 24881329
- [Background] Carbia C, Lannoy S, Maurage P, Lopez-Caneda E, O'Riordan KJ, Dinan TG, Cryan JF. A biological framework for emotional dysregulation in alcohol misuse: from gut to brain. Mol Psychiatry. 2021 Apr;26(4):1098-1118. doi: 10.1038/s41380-020-00970-6. Epub 2020 Dec 7. PMID 33288871
- [Background] Cryan JF, Dinan TG. Mind-altering microorganisms: the impact of the gut microbiota on brain and behaviour. Nat Rev Neurosci. 2012 Oct;13(10):701-12. doi: 10.1038/nrn3346. Epub 2012 Sep 12. PMID 22968153
- [Background] Cryan JF, O'Riordan KJ, Sandhu K, Peterson V, Dinan TG. The gut microbiome in neurological disorders. Lancet Neurol. 2020 Feb;19(2):179-194. doi: 10.1016/S1474-4422(19)30356-4. Epub 2019 Nov 18. PMID 31753762
- [Background] Leclercq S, Matamoros S, Cani PD, Neyrinck AM, Jamar F, Starkel P, Windey K, Tremaroli V, Backhed F, Verbeke K, de Timary P, Delzenne NM. Intestinal permeability, gut-bacterial dysbiosis, and behavioral markers of alcohol-dependence severity. Proc Natl Acad Sci U S A. 2014 Oct 21;111(42):E4485-93. doi: 10.1073/pnas.1415174111. Epub 2014 Oct 6. PMID 25288760
- [Background] Leclercq S, de Timary P, Delzenne NM, Starkel P. The link between inflammation, bugs, the intestine and the brain in alcohol dependence. Transl Psychiatry. 2017 Feb 28;7(2):e1048. doi: 10.1038/tp.2017.15. PMID 28244981
- [Background] Jadhav KS, Peterson VL, Halfon O, Ahern G, Fouhy F, Stanton C, Dinan TG, Cryan JF, Boutrel B. Gut microbiome correlates with altered striatal dopamine receptor expression in a model of compulsive alcohol seeking. Neuropharmacology. 2018 Oct;141:249-259. doi: 10.1016/j.neuropharm.2018.08.026. Epub 2018 Aug 31. PMID 30172845
- [Background] Leclercq S, Starkel P, Delzenne NM, de Timary P. The gut microbiota: A new target in the management of alcohol dependence? Alcohol. 2019 Feb;74:105-111. doi: 10.1016/j.alcohol.2018.03.005. Epub 2018 Mar 20. PMID 30031625
- [Background] Lannoy S, Billieux J, Dormal V, Maurage P. Behavioral and Cerebral Impairments Associated with Binge Drinking in Youth: A Critical Review. Psychol Belg. 2019 Mar 29;59(1):116-155. doi: 10.5334/pb.476. PMID 31328014
- [Background] Lopez-Caneda E, Crego A, Campos AD, Gonzalez-Villar A, Sampaio A. The Think/No-Think Alcohol Task: A New Paradigm for Assessing Memory Suppression in Alcohol-Related Contexts. Alcohol Clin Exp Res. 2019 Jan;43(1):36-47. doi: 10.1111/acer.13916. Epub 2018 Nov 25. PMID 30375668
- [Derived] Prata-Martins D, Nobre C, Almeida-Antunes N, Azevedo P, Sousa SS, Crego A, Cryan J, Sampaio A, Carbia C, Lopez-Caneda E. Assessing the impact of binge drinking and a prebiotic intervention on the gut-brain axis in young adults: protocol for a randomised controlled trial. BMJ Open. 2025 Sep 4;15(9):e095932. doi: 10.1136/bmjopen-2024-095932. PMID 40908013

DOCUMENTS (1):
  • Informed Consent Form (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT05946083/ICF_001.pdf